CLINICAL TRIAL: NCT01060319
Title: A Comprehensive Study to Isolate Tumor-initiating Cells From Human Epithelial Malignancies
Status: Withdrawn | Type: Observational
Why Stopped: Business Decision
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: BLDR0011; SU-11062009-4360 (Other: Stanford University)
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Bladder Cancer; Skin Cancers; Bladder (Urothelial, Transitional Cell) Cancer; Bladder (Urothelial, Transitional Cell) Cancer Resectable (Pre-Cystectomy)
MeSH Terms: conditions — Urinary Bladder Neoplasms; Skin Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bladder cancer specimens

SUMMARY:
We hypothesize that all human malignancies harbour a subpopulation of tumor initiating cells/cancer stem cells (CSCs) that drives tumor development and potentially recurrence or metastasis of the disease. The primary aim of this study is to develop strategies for prospective isolation/enrichment of CSCs from human tumors of different tissue origins. In addition, we will characterize the signaling pathways and/or tumor specific antigens that are specific for CSCs, in order to specifically target these CSCs as the endpoint of this study.

ELIGIBILITY:
Inclusion Criteria:N/A. We will recruit all non-melanoma skin and bladder cancer patients that are recommended for surgical removal of tumor tissues. This includes patients from all ages, gender and ethnicity background. Our sample collection criteria based on the tumor size of individual (e.g. tumor samples will only be collected if it will not affect the pathological diagnosis or treatment procedures of patients). Exclusion Criteria:N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-melanoma skin and bladder cancer patients that are recommended for surgical removal of tumor tissues
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of cancer stem cells (CSCs) | The current study does not include the active involvement of patients. Our study involves the collection of tumor samples from patients after surgical procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Irving L. Weissman M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States